CLINICAL TRIAL: NCT05427058
Title: Hypogastric Plexus Block and Ganglion Impar Block for Cervical and Endometrial Cancer Pain Management: A Randomized Controlled Trial of Efficacy and Safety
Brief Title: Hypogastric Plexus Block and Ganglion Impar Block for Cervical and Endometrial Cancer Pain Management
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Brawijaya (Other)
Responsible Party: Principal Investigator, Ristiawan Muji Laksono, MD, Principal Investigator, University of Brawijaya
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: UB_WWN01
Record Dates: First submitted 2022-03-29; First posted 2022-06-22 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Cervical Cancer; Endometrial Cancer
Keywords: Perineal Pain; Cervical Cancer; Endometrial Cancer; Superior Hypogastric Plexus Block; Ganglion Impar Block; pelvic pain
MeSH Terms: conditions — Uterine Cervical Neoplasms; Endometrial Neoplasms; Pelvic Pain

STUDY DESIGN:
Intervention Model Description: Patients were assigned to two groups.
  Group 1: Patients with pelvic floor pain due to cervical and endometrial cancer who were treated with superior hypogastric plexus block.
  Group 2: Patients with pelvic floor pain due to cervical and endometrial cancer who were given ganglion impar block.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant and Investigator masking:
  The random order of the groups will be written on paper and hidden by using a sealed envelope with consecutive numbers. This envelope will be retained by personnel who are not involved in the care or evaluation of the patient, or the analysis of the data.
  During the action, doctors and nurses are prohibited from communicating with participants regarding the actions given.
  Outcomes assessor masking:
  All data collection will be carried out by residents as research assistants who are trained for data collection. The assistant was not told what intervention was given to the patient, data collection was done directly by asking the patient without looking at the patient's status. The data that has been collected will be entered and processed by personnel outside the research team to ensure blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1: superior hypogastric plexus block group (Active Comparator): Device: C-arm fluoroscopic device Drug: lidocaine + alcohol
  Interventions: Procedure: Superior Hypogastric Plexus Block
- group 2: ganglion impar block group (Experimental): Device: C-arm fluoroscopic device Drug: lidocaine + alcohol
  Interventions: Procedure: Ganglion Impar Block

INTERVENTIONS:
Procedure: Superior Hypogastric Plexus Block — this procedure uses a transdiscal approach at the level of the L5-S1 vertebrae by injecting 5 ml of 1% lidocaine + 10 ml of 96% alcohol and confirmed by C-arm.
  Arms: group 1: superior hypogastric plexus block group
Procedure: Ganglion Impar Block — this procedure uses a trans-sacrococcygeal approach by injecting 4 ml of 1% lidocaine + 6 ml of 96% alcohol and confirmed by C-arm.
  Arms: group 2: ganglion impar block group

SUMMARY:
This study compared the efficacy and safety of superior hypogastric plexus block and ganglion impar block procedures on the management of pelvic and perineal cancer pain in patients with cervical and endometrial cancer

DETAILED DESCRIPTION:
Superior hypogastric plexus block is a commonly used method for the management of pelvic and perineal pain due to cancer, this procedure uses a transdiscal approach at the level of the L5-S1 vertebrae by injecting 5 ml of 1% lidocaine + 10 ml of 96% alcohol and confirmed by C-arm.

Compared with the ganglion impar block procedure using a trans-sacrococcygeal approach by injecting 4 ml of 1% lidocaine + 6 ml of 96% alcohol and confirmed by C-arm. The aim of this study was to compare the efficacy and safety of the ganglion impar block procedure against the superior hypogastric plexus block which is commonly used in the management of pelvic and perineal pain due to cervical and endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Unbearable cancer pain that is resistant to WHO (World Health Organization) pain ladder at least 2 weeks medication
* The patient is tired of taking medication orally or complications of current medication (respiratory depression, nausea, vomiting, opioid-induced constipation, gastrointestinal disturbances)
* Patients with pelvic floor pain diagnosed by a (Fellow of Interventional Pain Practice) FIPP-certified pain specialist
* Patients with pain in the perineum diagnosed by a FIPP-certified pain specialist
* Numerical Rating Scale >4
* >18 years old
* Able and willing to sign an informed consent

Exclusion Criteria:

* Refuse to be included in the research
* Blood clotting disorders (including taking anticoagulant drugs)
* Local infection in the area of action
* Loss to follow up

Drop-out Criteria:

* Loss to follow up
* Intervention complications occur
* Failed intervention

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Numerical rating scale (NRS) | 3 month
  Used to measure pain relief with a value of 0-10 (0 = no pain, 1-3 = mild pain, 4-6 = moderate pain, 7-9 = severe pain, 10 = most severe pain). The average pain intensity felt by the patient in the last 1 week
Oswestry Disability Index (ODI) | 3 Month
  The Oswestry Disability Index is a measuring tool to evaluate the quality of life and the level of disability. In this study, we will use the Indonesian adaptation version. in a journal published by Phedy et al showed that the Indonesian version of the ODI retains the reliability, validity, and psychometric characteristics of the original ODI.
  There are 10 main questions with 6 assessment options from the lowest point of 0 and the highest point of 5.
  0-20%: mild disability 21-40%: moderate disability, affecting activities can still be overcome 41-60%: severe disability, pain is a major problem and interferes with activities 61-80%: patients experience disturbances in major aspects of life requiring intervention 81-100%: the patient is confined to bed because of complaints
Morphine equivalent daily dose (MEDD) | 3 Month
  This is the dose that the patient takes regularly to relieve pain.

SECONDARY OUTCOMES:
Adverse effect | 3 Month
  It is an unwanted effect due to the intervention given to the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ristiawan M Laksono, Principal Investigator — Brawijaya University; Andika B Effendi, Study Director — Brawijaya University
Locations (1):
- General Hospital Saiful Anwar Malang, Malang, East Java, Indonesia

REFERENCES:
- [Background] Fowler JR, Maani EV, Dunton CJ, Gasalberti DP, Jack BW. Cervical Cancer. 2023 Nov 12. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK431093/ PMID 28613745
- [Background] Vrachnis N, Iavazzo C, Salakos N, Papamargaritis E, Boutas I, Creatsas G. Uterine tamponade balloon for the management of massive hemorrhage during cesarean section due to placenta previa/increta. Clin Exp Obstet Gynecol. 2012;39(2):255-7. PMID 22905480
- [Background] Yoon SY, Oh J. Neuropathic cancer pain: prevalence, pathophysiology, and management. Korean J Intern Med. 2018 Nov;33(6):1058-1069. doi: 10.3904/kjim.2018.162. Epub 2018 Jun 25. PMID 29929349
- [Background] Schmidt BL, Hamamoto DT, Simone DA, Wilcox GL. Mechanism of cancer pain. Mol Interv. 2010 Jun;10(3):164-78. doi: 10.1124/mi.10.3.7. PMID 20539035
- [Background] Bhatnagar S, Gupta M. Evidence-based Clinical Practice Guidelines for Interventional Pain Management in Cancer Pain. Indian J Palliat Care. 2015 May-Aug;21(2):137-47. doi: 10.4103/0973-1075.156466. PMID 26009665
- [Background] Gunduz OH, Kenis-Coskun O. Ganglion blocks as a treatment of pain: current perspectives. J Pain Res. 2017 Dec 14;10:2815-2826. doi: 10.2147/JPR.S134775. eCollection 2017. PMID 29276402
- [Background] Khan MA, Ashrafi SH, Decker SJ. The hepatic ultrastructure of chlordene-fed pigeons. Arch Environ Contam Toxicol. 1977;5(4):385-402. doi: 10.1007/BF02220919. PMID 196561
- [Background] Raja SN, Carr DB, Cohen M, Finnerup NB, Flor H, Gibson S, Keefe FJ, Mogil JS, Ringkamp M, Sluka KA, Song XJ, Stevens B, Sullivan MD, Tutelman PR, Ushida T, Vader K. The revised International Association for the Study of Pain definition of pain: concepts, challenges, and compromises. Pain. 2020 Sep 1;161(9):1976-1982. doi: 10.1097/j.pain.0000000000001939. PMID 32694387
- [Background] Tunio M, Al Asiri M, Bayoumi Y, Abdullah O Balbaid A, AlHameed M, Gabriela SL, Amir O Ali A. Lumbosacral plexus delineation, dose distribution, and its correlation with radiation-induced lumbosacral plexopathy in cervical cancer patients. Onco Targets Ther. 2014 Dec 23;8:21-7. doi: 10.2147/OTT.S71086. eCollection 2015. PMID 25565862
- [Background] Leslie KK, Thiel KW, Goodheart MJ, De Geest K, Jia Y, Yang S. Endometrial cancer. Obstet Gynecol Clin North Am. 2012 Jun;39(2):255-68. doi: 10.1016/j.ogc.2012.04.001. PMID 22640714
- [Background] Zhang S, Gong TT, Liu FH, Jiang YT, Sun H, Ma XX, Zhao YH, Wu QJ. Global, Regional, and National Burden of Endometrial Cancer, 1990-2017: Results From the Global Burden of Disease Study, 2017. Front Oncol. 2019 Dec 19;9:1440. doi: 10.3389/fonc.2019.01440. eCollection 2019. PMID 31921687
- [Background] Fallon MT. Neuropathic pain in cancer. Br J Anaesth. 2013 Jul;111(1):105-11. doi: 10.1093/bja/aet208. PMID 23794652
- [Background] Oliveira KG, von Zeidler SV, Podesta JR, Sena A, Souza ED, Lenzi J, Bissoli NS, Gouvea SA. Influence of pain severity on the quality of life in patients with head and neck cancer before antineoplastic therapy. BMC Cancer. 2014 Jan 24;14:39. doi: 10.1186/1471-2407-14-39. PMID 24460780
- [Background] van den Beuken-van Everdingen MH, de Graeff A, Jongen JL, Dijkstra D, Mostovaya I, Vissers KC; national guideline working group "Diagnosis treatment of cancer pain". Pharmacological Treatment of Pain in Cancer Patients: The Role of Adjuvant Analgesics, a Systematic Review. Pain Pract. 2017 Mar;17(3):409-419. doi: 10.1111/papr.12459. Epub 2016 May 21. PMID 27207115
- [Background] Hochberg U, Minerbi A, Boucher LM, Perez J. Interventional Pain Management for Cancer Pain: An Analysis of Outcomes and Predictors of Clinical Response. Pain Physician. 2020 Sep;23(5):E451-E460. PMID 32967396
- [Background] Ahmed DG, Mohamed MF, Mohamed SA. Superior hypogastric plexus combined with ganglion impar neurolytic blocks for pelvic and/or perineal cancer pain relief. Pain Physician. 2015 Jan-Feb;18(1):E49-56. PMID 25675070
- [Background] Schultz DM. Inferior hypogastric plexus blockade: a transsacral approach. Pain Physician. 2007 Nov;10(6):757-63. PMID 17987098
- [Background] Mohamed SA, Ahmed DG, Mohamad MF. Chemical neurolysis of the inferior hypogastric plexus for the treatment of cancer-related pelvic and perineal pain. Pain Res Manag. 2013 Sep-Oct;18(5):249-52. doi: 10.1155/2013/196561. Epub 2013 May 28. PMID 23717828
- [Background] Cariati M, De Martini G, Pretolesi F, Roy MT. CT-guided superior hypogastric plexus block. J Comput Assist Tomogr. 2002 May-Jun;26(3):428-31. doi: 10.1097/00004728-200205000-00019. PMID 12016374
- [Background] Turker G, Basagan-Mogol E, Gurbet A, Ozturk C, Uckunkaya N, Sahin S. A new technique for superior hypogastric plexus block: the posteromedian transdiscal approach. Tohoku J Exp Med. 2005 Jul;206(3):277-81. doi: 10.1620/tjem.206.277. PMID 15942158
- [Background] Gamal G, Helaly M, Labib YM. Superior hypogastric block: transdiscal versus classic posterior approach in pelvic cancer pain. Clin J Pain. 2006 Jul-Aug;22(6):544-7. doi: 10.1097/01.ajp.0000202978.06045.24. PMID 16788341
- [Background] Mishra S, Bhatnagar S, Gupta D, Thulkar S. Anterior ultrasound-guided superior hypogastric plexus neurolysis in pelvic cancer pain. Anaesth Intensive Care. 2008 Sep;36(5):732-5. doi: 10.1177/0310057X0803600518. PMID 18853596
- [Background] Jungquist CR, Vallerand AH, Sicoutris C, Kwon KN, Polomano RC. Assessing and Managing Acute Pain: A Call to Action. Am J Nurs. 2017 Mar;117(3 Suppl 1):S4-S11. doi: 10.1097/01.NAJ.0000513526.33816.0e. PMID 28212145
- [Background] Swieboda P, Filip R, Prystupa A, Drozd M. Assessment of pain: types, mechanism and treatment. Ann Agric Environ Med. 2013;Spec no. 1:2-7. PMID 25000833
- [Background] Nicholas M, Vlaeyen JWS, Rief W, Barke A, Aziz Q, Benoliel R, Cohen M, Evers S, Giamberardino MA, Goebel A, Korwisi B, Perrot S, Svensson P, Wang SJ, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic primary pain. Pain. 2019 Jan;160(1):28-37. doi: 10.1097/j.pain.0000000000001390. PMID 30586068
- [Background] Treede RD, Rief W, Barke A, Aziz Q, Bennett MI, Benoliel R, Cohen M, Evers S, Finnerup NB, First MB, Giamberardino MA, Kaasa S, Korwisi B, Kosek E, Lavand'homme P, Nicholas M, Perrot S, Scholz J, Schug S, Smith BH, Svensson P, Vlaeyen JWS, Wang SJ. Chronic pain as a symptom or a disease: the IASP Classification of Chronic Pain for the International Classification of Diseases (ICD-11). Pain. 2019 Jan;160(1):19-27. doi: 10.1097/j.pain.0000000000001384. PMID 30586067
- [Background] Colloca L, Ludman T, Bouhassira D, Baron R, Dickenson AH, Yarnitsky D, Freeman R, Truini A, Attal N, Finnerup NB, Eccleston C, Kalso E, Bennett DL, Dworkin RH, Raja SN. Neuropathic pain. Nat Rev Dis Primers. 2017 Feb 16;3:17002. doi: 10.1038/nrdp.2017.2. PMID 28205574
- [Background] Yoo SK, Starnes TW, Deng Q, Huttenlocher A. Lyn is a redox sensor that mediates leukocyte wound attraction in vivo. Nature. 2011 Nov 20;480(7375):109-12. doi: 10.1038/nature10632. PMID 22101434
- [Background] Falk S, Dickenson AH. Pain and nociception: mechanisms of cancer-induced bone pain. J Clin Oncol. 2014 Jun 1;32(16):1647-54. doi: 10.1200/JCO.2013.51.7219. Epub 2014 May 5. PMID 24799469
- [Background] Davis MP. Drug management of visceral pain: concepts from basic research. Pain Res Treat. 2012;2012:265605. doi: 10.1155/2012/265605. Epub 2012 Apr 24. PMID 22619712
- [Background] Yam MF, Loh YC, Tan CS, Khadijah Adam S, Abdul Manan N, Basir R. General Pathways of Pain Sensation and the Major Neurotransmitters Involved in Pain Regulation. Int J Mol Sci. 2018 Jul 24;19(8):2164. doi: 10.3390/ijms19082164. PMID 30042373
- [Background] Lema MJ, Foley KM, Hausheer FH. Types and epidemiology of cancer-related neuropathic pain: the intersection of cancer pain and neuropathic pain. Oncologist. 2010;15 Suppl 2:3-8. doi: 10.1634/theoncologist.2009-S505. PMID 20489190
- [Background] Starobova H, Vetter I. Pathophysiology of Chemotherapy-Induced Peripheral Neuropathy. Front Mol Neurosci. 2017 May 31;10:174. doi: 10.3389/fnmol.2017.00174. eCollection 2017. PMID 28620280
- [Background] van den Beuken-van Everdingen MH, Hochstenbach LM, Joosten EA, Tjan-Heijnen VC, Janssen DJ. Update on Prevalence of Pain in Patients With Cancer: Systematic Review and Meta-Analysis. J Pain Symptom Manage. 2016 Jun;51(6):1070-1090.e9. doi: 10.1016/j.jpainsymman.2015.12.340. Epub 2016 Apr 23. PMID 27112310
- [Background] Baldini A, Von Korff M, Lin EH. A Review of Potential Adverse Effects of Long-Term Opioid Therapy: A Practitioner's Guide. Prim Care Companion CNS Disord. 2012;14(3):PCC.11m01326. doi: 10.4088/PCC.11m01326. Epub 2012 Jun 14. PMID 23106029
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Prabhu M, Eckert LO. Development of World Health Organization (WHO) recommendations for appropriate clinical trial endpoints for next-generation Human Papillomavirus (HPV) vaccines. Papillomavirus Res. 2016 Dec;2:185-189. doi: 10.1016/j.pvr.2016.10.002. Epub 2016 Oct 26. PMID 29074180
- [Background] Rocha A, Plancarte R, Nataren RGR, Carrera IHS, Pacheco VALR, Hernandez-Porras BC. Effectiveness of Superior Hypogastric Plexus Neurolysis for Pelvic Cancer Pain. Pain Physician. 2020 Mar;23(2):203-208. PMID 32214302
- [Background] Gonnade N, Mehta N, Khera PS, Kumar D, Rajagopal R, Sharma PK. Ganglion impar block in patients with chronic coccydynia. Indian J Radiol Imaging. 2017 Jul-Sep;27(3):324-328. doi: 10.4103/ijri.IJRI_294_16. PMID 29089683
- [Background] Bakshi SG, Rathod A, Salunkhe S. Influence of interpretation of pain scores on patients' perception of pain: A prospective study. Indian J Anaesth. 2021 Mar;65(3):216-220. doi: 10.4103/ija.IJA_130_21. Epub 2021 Mar 13. PMID 33776112
- [Background] Phedy P, Djaja YP, Tobing SDAL, Gatam L, Librianto D, Fachrisal, Gatam AR, Hardiansyah NP. Cross-cultural adaptation and psychometric validation of the Indonesian version of the Oswestry Disability Index. Eur Spine J. 2021 Apr;30(4):1053-1062. doi: 10.1007/s00586-020-06690-3. Epub 2021 Jan 2. PMID 33389199
- [Background] Bhatnagar S, Khanna S, Roshni S, Goyal GN, Mishra S, Rana SP, Thulkar S. Early ultrasound-guided neurolysis for pain management in gastrointestinal and pelvic malignancies: an observational study in a tertiary care center of urban India. Pain Pract. 2012 Jan;12(1):23-32. doi: 10.1111/j.1533-2500.2011.00467.x. Epub 2011 May 26. PMID 21615855